CLINICAL TRIAL: NCT07087964
Title: Positron Emission Tomography With Innovative Laboratory Techniques for Improved Risk and Disease Assessment in Myeloma
Brief Title: Positron Emission Tomography With Innovative Laboratory Techniques for Improved Risk and Disease Assessment in Newly Diagnosed Multiple Myeloma Patients
Acronym: IMMPROVED
Status: Recruiting | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: FWO Research Fund Flanders (Unknown); Universitaire Ziekenhuizen KU Leuven (Other); University Ghent (Other); University Hospital, Antwerp (Other); Amsterdam UMC, location VUmc (Other); AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sébastien Anguille, Prof. Dr., Universiteit Antwerpen
Other Study IDs: FWO-TBM T003420N; 2021-005864-22 (EudraCT Number)
Record Dates: First submitted 2025-06-25; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Newly Diagnosed Multiple Myeloma (NDMM)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At diagnosis (and in case of relapse): if possible an additional bone marrow aspirate sample will be taken during a routine investigation. This sample will be processed for whole exome sequencing (WES). This is a genetic test performed with the aim to gain more information on the genetic background of the disease. The samples will be completely used and will not be stored after end of study.
  All the other samples taken are part of standard of care and hospital policy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed Mulitple myeloma (NDMM) patients: Patients who recently received the diagnosis multiple myeloma and who will start a standard of care treatment consisting of induction chemotherapy and autologous stem cell transplantation (ASCT), followed by maintenance therapy.
  If a patient has already started therapy, it is still possible to be included in the study if following conditions are met: whole body FDG PET/LDCT scan at diagnosis and obtaining at least a very good partial response (VGPR) before start of maintenance therapy.

SUMMARY:
This study investigates newly diagnosed multiple myeloma patients following standard of care treatment. The primary endpoint of the study is to determine minimal residual disease (MRD) by combining 2 techniques in order to better predict progression free survival (PFS) of a patient. Secondary endpoint is to gain more insight into diagnostic features to better stratify patients based on risk factors for early relapse. Both endpoints could lead to a more patient specific treatment in the future.

Participants will be followed throughout their standard of care treatment. This treatment consists of indcution chemotherapy, followed by autologous stem cell transplant (ASCT), followed by lenalidomide maintenance therapy.

* Before start of induction chemotherapy the patient will receive a whole-body FDG PET/LDCT scan and an additional bone marrow aspirate sample will be taken during a routine bone marrow punction. This sample will be used for whole exome sequencing (WES).
* For those patients who achieve at least a very good partial response (VGPR) after induction chemotherapy and ASCT a repeat whole body FDG PET/LDCT scan will be performed before start of maintenance therapy. This scan will be repeated for a third time after 1 year of maintenance therapy. Besides this, an additional bone marrow aspirate sample will be taken for MRD detection. This will be done before start of maintenance therapy, after 1 year of maintenance therapy and after 2 years of maintenance therapy. MRD detection is done by next generation flow cytometery (NGF).
* During mantenance therapy patient follow-up will be performed at least every 3 months to determine best response to therapy or possible relapse (based on routine lab information).
* Those patients who do not achieve VGPR or better will not need to receive a whole body FDG PET/CT scan and MRD detection by flow cytometry, but these patients will undergo the same follow-up during maintenance therapy.
* In case of relapse, for all patients, an additional bone marrow aspirate sample will be taken for WES (during a routine bone marrow investigation).

ELIGIBILITY:
Inclusion Criteria:

* Transplant-eligible newly diagnosed multiple myeloma based on current IMWG criteria and scheduled for induction chemotherapy followed by ASCT. Remark: patiënts can also be included after ASCT, prior to maintenance therapy, if a baseline FDG-PET CT scan showing FDG avid disease is available.
* Baseline 18F-FDG PET/WBLDCT scan should be performed before start of treatment (preferably) or within 7 days after start of treatment. Scan must show FDG avid disease (=at least 1 FL ≥ DS3 and/or diffuse bone marrow involvement).
* WHO performance status 0-2 (WHO > 2 can be allowed if due to underlying disease and after discussion with the physician).
* Age ≥ 18 years
* Life expectancy > 12 months, based on clinical judgement.

Eligibility criteria for the primary endpoint

* achieving at least a VGPR after induction chemotherapy and ASCT according to the standard IMWG response criteria.
* received at least one (28-day) cycle of lenalidomide as maintenance therapy after ASCT. No new therapy can be given until clinical relapse.

Exclusion Criteria:

* Any physical or physiological condition that may affect adherence to the study protocol, e.g. severe claustrophobia or the inability to lie still for 30 minutes.
* uncontrolled diabetes
* History of concomitant presence of any other malignancy, except for:

  * non-melanoma skin cancer
  * carinoma in situ of the cervix
  * any other effectively treated malignancy that has been in remission for > 5 years or that is highly likely to be cured at the time of enrollment.
* pregnant or breastfeeding
* refusal or inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed multiple myeloma patients will be included at participating centers: Universitair ziekenhuis Antwerpen, Universitair Ziekenhuis Gent, Universitair Ziekenhuis Leuven, AZ Sint-Jan Brugge and UMC Amsterdam (the Netherlands).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of MRD assessment by FDG-PET combined with NGF in patiënts achieving VGPR or better after induction chemotherapy and ASCT | From achieving VGPR and measuring MRD by FDG PET/CT and NGF until the patiënt received 2 years of maintenance therapy (or until detection of progressive disease or dead, whichever occurs first).
  The investigators hypothesize that only patients who have no evidence of disease on both NGF and FDG-PET (MRD double negative) have a durable response with a 2y PFS of 90% compared to 50% in patients who have evidence of disease on at least one modality (MRD positive).
  PFS is defined as the time from achieving ≥ VGPR and confirmation of absence of MRD (landmark) to first documentation of objective progressive disease or death due to any cause, whichever occurs first.
  The <10^-5 MRD level is used to define BM-NGF MRD negativity. A Deauville score = 3 threshold will be used to define FDG-PET MRD negativity, but alternatives will also be evaluated (other DS, more quantitative measures like SUV).

SECONDARY OUTCOMES:
Improvement of risk stratification at baseline - based on WES | From diagnosis until progression, death or end of follow-up period (2years of maintenance therapy).
  The secondary endpoint is to implement WES and Radiomics at baseline to improve risk-stratification. Looking at WES-analysis: WES at baseline will be correlated with PFS duration, in order to explore wether certain WES signatures are correlated with shorter or longer PFS.
Improvement of risk stratification at baseline - based on radiomics | From diagnosis until progression, death or end of follow-up period (2years of maintenance therapy).
  The secondary endpoint is to implement WES and Radiomics at baseline to improve risk-stratification. Lookting at radiomics: PET radiomics will be perforemd and correlated with PFS duration. Is there a significant difference (higher/lower) between patients with a PFS of >24 months vs patients who show PD during maintenance therapy (PFS < 24 months).

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - Universitair ziekenhuis Antwerpen, Antwerp, Antwerpen
  - Universitair ziekenhuis Gent, Ghent, Oost Vlaandere
  - Universitair Ziekenhuis Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge, Bruges, West-Vlaandere